CLINICAL TRIAL: NCT04000997
Title: The Predictive Value of Cough Peak Flow for Extubation Success in Mechanically Ventilated Patients After Craniotomy: a Single-center Prospective Diagnostic Study
Brief Title: The Predictive Value of Peak Cough Flow for Endotracheal Extubation of Patients After Craniotomy
Acronym: PCFET
Status: Completed | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Jianfang Zhou, MD, Beijing Tiantan Hospital
Other Study IDs: JZhou-1
Record Dates: First submitted 2019-06-26; First posted 2019-06-27 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-02

CONDITIONS: Extubation Success; Craniofacial Pain Syndrome; Cough Peak Flow; Endotracheal Tube
Keywords: endotracheal tube; extubation success; cough peak flow; predictive value; post-craniotomy; critically ill
MeSH Terms: conditions — Facial Neuralgia; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Failure group: Patients with a failure extubation
- Success group: Patients with a successful extubation

SUMMARY:
In severe cases after craniotomy, tracheal intubation is often required, and the removal of tracheal intubation presents certain risks and challenges. Premature removal of the tracheal intubation can lead to failure of extubation and increased proportion of re-intubation, resulting in increased risk of airway injury and hospital-acquired pneumonia, resulting in prolonged hospital stay and even adverse effects on neurological outcomes and mortality. However, delayed extubation can also lead to an increased risk of hospital acquired pneumonia, affecting early recovery and neurological recovery. It can be seen that the accurate evaluation of the possibility of tracheal intubation and the appropriate timing can have a greater impact on the prognosis of patients after craniotomy. However, there are currently no relevant standards or guidelines to guide clinical work. Previous studies have shown that for general critically ill patients, Peak cough flow (PCF) can play a certain role in predicting tracheal intubation, but the results of each study are not consistent. The predictive value of PCF for tracheal intubation and extubation in patients after craniotomy is less relevant. This study intends to use Pneumotachograph to measure the active and passive PCF of patients with extubation, to explore the predictive value of PCF for tracheal intubation after craniotomy, and to provide guidance for the development of clinical extubation decisions.

DETAILED DESCRIPTION:
The objection of this study is to evaluate the preditive value of PCF for endotracheal extubation in patients undergoing craniotomy. For patients who met the inclusion criteria, the PCF value will be measured before the removal of entracheal tubes, and the predictive value of PCF will be evaluated by ROC curves, as will as the cut-off value of PCF.

According to state of consciousness, patients will be grouped as consciousness and unconsciousness group, and the predictive value of PCF for endotracheal extubation will be evaluated seprately in both groups. For patients with disturbance of consciousness, only passive PCF value will be measured. For lucid patients, inaddition to passive PCF value, the voluntary PCF value will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Post- craniotomy
* ICU LOS ≥ 24h

Exclusion Criteria:

* no extubation attempt during the ICU stay;
* underwent tracheostomy without extubation attempt;
* pregnant or lactating women;
* enrolled in other clinical trials;
* declined to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted into ICU ward after craniotomy will be screened. Those ones meeting the including criteria will be included. patients would be grouped by their extubation outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 785 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Predictive value of CPF for endotracheal extubation | 72h after extubation
  Failure of extubation refers to re-intubation within 72 hours after extubation

SECONDARY OUTCOMES:
mortality rates | in hospital
  Comparison of mortality rates between patients with failed extubation and successful extubation.

CONTACTS AND LOCATIONS:
Overall Officials: Jianxin Zhou, MD, Study Director — Beijing Tian Tan Hospital
Locations (1):
- Jianfang Zhou, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Data sets generated during the current study are available from the first author on reasonable request.
Supporting Information: SAP
Time Frame: June to December 2025
Access Criteria: It is necessary to provide materials related to the purpose of the data and the usage plan, and sign a data sharing agreement. In addition, the use of the data is subject to the approval of the Ethics Committee of our hospital. The first author can be contacted by email.

REFERENCES:
- [Background] Reis HF, Almeida ML, Silva MF, Rocha Mde S. Extubation failure influences clinical and functional outcomes in patients with traumatic brain injury. J Bras Pneumol. 2013 May-Jun;39(3):330-8. doi: 10.1590/S1806-37132013000300010. PMID 23857695
- [Background] McCredie VA, Ferguson ND, Pinto RL, Adhikari NK, Fowler RA, Chapman MG, Burrell A, Baker AJ, Cook DJ, Meade MO, Scales DC; Canadian Critical Care Trials Group. Airway Management Strategies for Brain-injured Patients Meeting Standard Criteria to Consider Extubation. A Prospective Cohort Study. Ann Am Thorac Soc. 2017 Jan;14(1):85-93. doi: 10.1513/AnnalsATS.201608-620OC. PMID 27870576
- [Background] Hyde GA, Savage SA, Zarzaur BL, Hart-Hyde JE, Schaefer CB, Croce MA, Fabian TC. Early tracheostomy in trauma patients saves time and money. Injury. 2015 Jan;46(1):110-4. doi: 10.1016/j.injury.2014.08.049. Epub 2014 Sep 16. PMID 25441577
- [Background] Alali AS, Scales DC, Fowler RA, Mainprize TG, Ray JG, Kiss A, de Mestral C, Nathens AB. Tracheostomy timing in traumatic brain injury: a propensity-matched cohort study. J Trauma Acute Care Surg. 2014 Jan;76(1):70-6; discussion 76-8. doi: 10.1097/TA.0b013e3182a8fd6a. PMID 24368359
- [Background] Bosel J, Schiller P, Hook Y, Andes M, Neumann JO, Poli S, Amiri H, Schonenberger S, Peng Z, Unterberg A, Hacke W, Steiner T. Stroke-related Early Tracheostomy versus Prolonged Orotracheal Intubation in Neurocritical Care Trial (SETPOINT): a randomized pilot trial. Stroke. 2013 Jan;44(1):21-8. doi: 10.1161/STROKEAHA.112.669895. Epub 2012 Nov 29. PMID 23204058
- [Background] Herritt B, Chaudhuri D, Thavorn K, Kubelik D, Kyeremanteng K. Early vs. late tracheostomy in intensive care settings: Impact on ICU and hospital costs. J Crit Care. 2018 Apr;44:285-288. doi: 10.1016/j.jcrc.2017.11.037. Epub 2017 Dec 22. PMID 29223743
- [Background] Kaese S, Zander MC, Lebiedz P. Successful Use of Early Percutaneous Dilatational Tracheotomy and the No Sedation Concept in Respiratory Failure in Critically Ill Obese Subjects. Respir Care. 2016 May;61(5):615-20. doi: 10.4187/respcare.04333. Epub 2016 Jan 12. PMID 26759420
- [Background] Wang R, Pan C, Wang X, Xu F, Jiang S, Li M. The impact of tracheotomy timing in critically ill patients undergoing mechanical ventilation: A meta-analysis of randomized controlled clinical trials with trial sequential analysis. Heart Lung. 2019 Jan;48(1):46-54. doi: 10.1016/j.hrtlng.2018.09.005. Epub 2018 Oct 15. PMID 30336945
- [Background] Tipping CJ, Harrold M, Holland A, Romero L, Nisbet T, Hodgson CL. The effects of active mobilisation and rehabilitation in ICU on mortality and function: a systematic review. Intensive Care Med. 2017 Feb;43(2):171-183. doi: 10.1007/s00134-016-4612-0. Epub 2016 Nov 18. PMID 27864615
- [Background] Pisegna JM, Murray J. Clinical Application of Flexible Endoscopic Evaluation of Swallowing in Stroke. Semin Speech Lang. 2018 Feb;39(1):3-14. doi: 10.1055/s-0037-1608855. Epub 2018 Jan 22. PMID 29359301
- [Derived] Zhou J, Li HL, Luo XY, Chen GQ, Yang YL, Zhang L, Xu M, Shi GZ, Zhou JX. Predictive value of cough peak flow for successful extubation in mechanically ventilated patients after craniotomy: a single-centre prospective diagnostic study. BMJ Open. 2025 Jan 2;15(1):e088219. doi: 10.1136/bmjopen-2024-088219. PMID 39753249